CLINICAL TRIAL: NCT01955434
Title: Phase II Study of LCL161 Alone and in Combination With Cyclophosphamide in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: SMAC Mimetic LCL161 Alone or With Cyclophosphamide in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1381; NCI-2013-01276 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CLCL161AUS01T; MC1381 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2016-08

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; LCL161

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (SMAC mimetic LCL161 and cyclophosphamide) (Experimental): Patients receive SMAC mimetic LCL161 PO QD on days 1, 8, 15, and 22. Patients lacking a minor response by end of course 2 or partial response by end of course 4 may also receive cyclophosphamide PO QD on days 1, 8, 15, and 22 at the discretion of the treating physician. Patients taking cyclophosphamide with less than a 25% interval reduction in paraprotein receive SMAC mimetic LCL161 on days 2, 9, 16, and 23. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Drug: Smac Mimetic LCL161

INTERVENTIONS:
Drug: Cyclophosphamide — Given PO
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Smac Mimetic LCL161 — Given PO
  Other Names: LCL161

SUMMARY:
This phase II trial studies how well second mitochondrial-derived activator of caspases (SMAC) mimetic LCL161 alone or with cyclophosphamide works in treating patients with multiple myeloma that has returned or does not respond to treatment. Biological therapies, such as SMAC mimetic LCL161, may stimulate the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving SMAC mimetic LCL161 alone or with cyclophosphamide is more effective in treating multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the confirmed overall response rate (>= partial response [PR]) to LCL161 (SMAC mimetic LCL161), used as a single agent, in patients with relapsed multiple myeloma (MM).

SECONDARY OBJECTIVES:

I. To estimate the confirmed overall response rate to LCL161 in combination with cyclophosphamide, when cyclophosphamide is added to LCL161 for lack of response or progression.

II. To estimate the overall survival and event-free survival of patients treated with LCL161 in combination with cyclophosphamide, when cyclophosphamide is added to LCL161 for lack of response or progression.

III. To evaluate the tolerability of LCL161 alone and in combination with cyclophosphamide in patients with relapsed MM.

TERTIARY OBJECTIVES:

I. To determine degradation of cellular inhibitor of apoptosis protein-1 (cIAP1) in peripheral blood mononuclear cells (PBMC), changes in serum cytokines, and changes in immune cell subsets by flow cytometry.

II. To correlate the effect of LCL161 with the presence of activating mutations of the nuclear factor kappa beta (NFKB) pathway.

III. To evaluate the pharmacokinetics (PK) of LCL161 alone, and LCL161 in combination with cyclophosphamide.

IV. To describe patient-reported health-related quality of life and symptoms.

OUTLINE:

Patients receive SMAC mimetic LCL161 orally (PO) once daily (QD) on days 1, 8, 15, and 22. Patients lacking a minor response by end of course 2 or partial response by end of course 4 may also receive cyclophosphamide PO QD on days 1, 8, 15, and 22 at the discretion of the treating physician. Patients taking cyclophosphamide with less than a 25% interval reduction in paraprotein receive SMAC mimetic LCL161 on days 2, 9, 16, and 23. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory multiple myeloma and has already received =< 4 standard treatment regimens; note: induction, transplant, consolidation, and maintenance is considered one regimen
* Have received prior therapy with an immunomodulatory agent, a proteosome inhibitor, and glucocorticoids
* Absolute neutrophil count (ANC) >= 1000/uL
* Untransfused platelet count >= 75,000/uL
* Aspartate aminotransferase (AST) =< 3 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) =< 3 x ULN
* Total bilirubin =< 1.5 mg/dL
* Serum creatinine =< 2.5 mg/dL
* Hemoglobin >= 8 g/dL
* Measurable disease of multiple myeloma as defined by at least ONE of the following:

  * Serum monoclonal protein >= 1.0 g/dL
  * >= 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * Monoclonal plasmacytosis >= 30% (evaluable disease)
  * Measurable plasmacytoma that has not been radiated
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, 2
* Willing and able to comply with scheduled visits, treatment plan and laboratory tests
* Able to swallow and retain oral medication
* Provide informed written consent
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Willing to provide all biological specimens as required by the protocol for correlative research purposes
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Mayo Clinic Arizona only: Willing to participate in associated biobanking study, 919-04; the patient must sign consent to enroll onto the mandatory companion biobanking study in order to participate in this treatment study
* Mayo Clinic Rochester and Florida only: Willing to participate in associated biobanking study, 521-93; the patient must sign consent to enroll onto the mandatory companion biobanking study in order to participate in this treatment study

Exclusion Criteria:

* Prior use of investigational drugs =< 14 days prior to registration
* Prior use of growth factors =< 14 days prior to registration
* Prior radiation therapy =< 14 days prior to registration
* Prior autologous stem cell transplant =< 12 weeks prior to registration
* Any of the following:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential who are unwilling to employ adequate contraception while receiving treatment on this study and for 4 months after stopping treatment on this study
  * Men who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while receiving treatment on this study and for 4 months after stopping treatment on this study NOTE: Postmenopausal women are allowed to participate in this study; women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago; in the case of oophorectomy alone, a woman is considered to be of not child bearing potential only when her reproductive status has been confirmed by follow-up hormone level assessment
* Prior allogeneic transplant of any kind
* Known active infection requiring parenteral or oral anti-infective treatment
* Serious psychiatric illness, active alcoholism, or drug addiction that may hinder or confuse follow-up evaluation
* Known human immunodeficiency virus (HIV) or active hepatitis B or C viral infection
* Active autoimmune/inflammatory conditions requiring ongoing immunosuppressive therapy
* Use of more than low dose corticosteroids (e.g., prednisone up to but no more than 10 mg PO QD or its equivalent) for symptom management and comorbid conditions, except for the following:

  * Topical applications (e.g. rash)
  * Inhaled sprays (e.g. obstructive airways diseases)
  * Eye drops or local injections (e.g. intra-articular)
  * Joint injections (e.g. arthritis) Doses of corticosteroid should be stable for at least 7 days prior to registration
* Any concurrent severe and/or uncontrolled medical conditions that could increase the patient's risk for toxicity while in the study or that could confound discrimination between disease- and study treatment-related toxicities
* Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

  * History or presence of ventricular tachyarrhythmia
  * Presence of unstable atrial fibrillation (ventricular response > 100 bpm) (NOTE: patients with stable atrial fibrillation are eligible, provided they do not meet any of the other cardiac exclusion criteria)
  * Clinically significant resting bradycardia (< 50 bpm)
  * Angina pectoris or acute myocardial infarction =< 3 months prior to registration
  * Other clinically significant heart disease (e.g., symptomatic congestive heart failure; uncontrolled arrhythmia or hypertension; history of labile hypertension or poor compliance with an antihypertensive regimen)
* Currently receiving treatment with agents that are metabolized solely through cytochrome P450, family 3, subfamily A, polypeptide 4/5 (CYP3A4/5) and have a narrow therapeutic index or are strong cytochrome P450, family 2, subfamily C, polypeptide 8 (CYP2C8) inhibitors; or are receiving treatment with agents that carry a risk for QT prolongation and are CYP3A substrates; caution should be used in patients taking other CYP2C8- or CYP3A4/5-interacting agents
* Impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of LCL161

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-11; Primary Completion 2016-06-09 (Actual); Study Completion 2016-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bergsagel, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (SMAC Mimetic LCL161 and Cyclophosphamide): Patients receive SMAC mimetic LCL161 (1200 mg) PO QD on days 1, 8, 15, and 22. Patients lacking a minor response by end of course 2 or partial response by end of course 4 may also receive cyclophosphamide (500 mg) PO QD on days 1, 8, 15, and 22 at the discretion of the treating physician. Patients taking cyclophosphamide with less than a 25% interval reduction in paraprotein receive SMAC mimetic LCL161 on days 2, 9, 16, and 23. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (SMAC Mimetic LCL161 and Cyclophosphamide)
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (SMAC Mimetic LCL161 and Cyclophosphamide)
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 68.0 [47.0 to 90.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Overall Response Rate (Stringent Complete Response [sCR], Complete Response [CR], Very Good Partial Response [VGPR], or Partial Response [PR]) With Single Agent SMAC Mimetic LCL161
Description: The primary endpoint of this study is the confirmed overall response rate with single agent LCL161 (prior to initiation of cyclophosphamide). A confirmed overall response is defined as sCR (CR as defined+Normal FLC ratio+Absence of clonal PCs by immunohistochemistry), CR (Negative immunofixation of serum and urine+Disappearance of any soft tissue plasmacytoma+<5% PCs in Bone Marrow+a normal FLC ratio), VGPR (Serum and urine M-component detectable by immunofixation but not on electrophoresis), or PR (If present at baseline, ≥ 50% reduction of serum M-protein and reduction in 24-hour urinary M-protein or to <200 mg/24hrs) noted as the objective status on two consecutive evaluations while receiving single agent LCL161.The rate (percentage) of successes will be estimated by the number of successes divided by the total number of evaluable patients times 100. 95% confidence intervals for the true success percentage will be calculated by the exact binomial method.
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (SMAC Mimetic LCL161 and Cyclophosphamide)
Number analyzed (Participants) | 25
percentage of patients | 0 [0 to 13.7]

2. Secondary Outcome: Combination Agent Response Rate
Description: The overall response rate (percentage) with the addition of cyclophosphamide will be estimated by the number of patients who achieve a confirmed overall response at any time (with SMAC mimetic LCL161 plus cyclophosphamide) divided by the number of evaluable patients times 100. 95% confidence intervals for the true confirmed overall response rate will be calculated by the exact binomial method.
Time Frame: Up to 1 year
Population: Patients treated with combination of LCL161 and cyclophosphamide were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (SMAC Mimetic LCL161 and Cyclophosphamide)
Number analyzed (Participants) | 23
percentage of patients | 17.4 [5.0 to 38.8]

3. Secondary Outcome: Event-free Survival
Description: The event-free survival time is defined as the time from registration to disease progression while receiving LCL161 and cyclophosphamide, death due to any cause, or subsequent treatment for multiple myeloma. Date of progression will be defined as the date that the criteria for progressive disease were first met after initiation of cyclophosphamide. If a patient goes off study treatment and never received cyclophosphamide, they will be censored on the date they went off study treatment. If a patient initiates cyclophosphamide but later discontinues cyclophosphamide due to toxicity and continues LCL161 alone, disease progression on LCL161 alone will be considered an event in this case. The distribution of event-free survival will be estimated using the method of Kaplan-Meier.
Time Frame: From registration to disease progression while receiving SMAC mimetic LCL161 and cyclophosphamide, death due to any cause, or subsequent treatment for multiple myeloma, assessed up to 1 year
Population: Patients treated with combination of LCL161 and cyclophosphamide were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (SMAC Mimetic LCL161 and Cyclophosphamide)
Number analyzed (Participants) | 23
months | 10.0 [4.6 to 24.4]

4. Secondary Outcome: Incidence of Toxicities Graded Using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 (All Treatment)
Description: The maximum grade for each type of adverse event, regardless of causality, will be recorded and reported for each patient, and frequency tables will be reviewed to determine adverse event patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. The percentage of patients with a maximum grade 3 or higher adverse event are reported below.
Time Frame: Up to 30 days after the last day of study drug treatment
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (SMAC Mimetic LCL161 and Cyclophosphamide)
Number analyzed (Participants) | 25
percentage of patients
  Anemia | 24
  Fatigue | 16
  Nausea | 4.0
  Platelet count decreased | 12.0
  Neutrophil count decreased | 36.0
  Lymphocyte count decreased | 52.0
  Vomiting | 4.0
  White blood cell decreased | 20.0
  Diarrhea | 4.0
  Rash maculo-papular | 4.0
  Hyperglycemia | 12.0
  Lymphocyte count increased | 8
  Syncope | 12.0
  Hyperuricemia | 4.0
  Hypotension | 4.0
  Lung infection | 4.0
  Pain in extremity | 4.0
  Sepsis | 4.0
  Uriticaria | 4.0

5. Secondary Outcome: Overall Survival
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: From registration to death due to any cause, assessed up to 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (SMAC Mimetic LCL161 and Cyclophosphamide)
Number analyzed (Participants) | 25
months | NA [NA to NA] — The median overall survival was not reached, and the lower and upper limits of the 95% confidence interval were not available.

6. Other Pre Specified Outcome: Activating Mutations of the NFKB Pathway
Description: Continuous biomarker levels will be explored in a graphical manner including mean plots and plots of change and percent change from baseline and other summary measures. Any potential relationships between the baseline level or change in the level of each biomarker and clinical outcome such as confirmed overall response, 6-month progression-free survival, and adverse event incidence will be further analyzed using Wilcoxon rank sum tests or logistic regression methods, as appropriate. Association between a mutation status and confirmed overall response will be assessed using a chi-squared test.
Time Frame: Up to 1 year
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Patient-reported Outcomes (Quality of Life and Symptoms)
Description: Scale score trajectories over time will be examined using stream plots and mean plots with standard deviation error bars overall. Changes from baseline at each cycle will be statistically tested using paired t-tests, and standardized response means (mean of the change from baseline scores at a given cycle, divided by the standard deviation of the change scores) will be interpreted (after applying Middel's adjustment) using Cohen's cut-offs. Correlation between outcomes will employ Pearson and/or Spearman correlations at individual time points.
Time Frame: Baseline up to 1 year
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Changes in Immune Cell Subsets
Description: as for outcome 6
Time Frame: Baseline up to 1 year
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Changes in Serum Cytokines
Description: as for outcome 6
Time Frame: Baseline up to 1 year
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Degradation of cIAP1 in PBMC
Description: as for outcome 6
Time Frame: Baseline up to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From baseline up to 30 days after last dose of study treatment
Description: CTCAE term (AE description) and grade: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. Each CTCAE term in the current version is a unique representation of a specific event used for medical documentation and scientific analysis and is a single MedDRA Lowest Level Term (LLT)
Arm/Group | Treatment (SMAC Mimetic LCL161 and Cyclophosphamide)
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 11/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (SMAC Mimetic LCL161 and Cyclophosphamide) (N=25)
Cytokine release syndrome (Immune system disorders) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (SMAC Mimetic LCL161 and Cyclophosphamide) (N=25)
Anemia (Blood and lymphatic system disorders) | 24 (133)
Abdominal pain (Gastrointestinal disorders) | 6 (16)
Constipation (Gastrointestinal disorders) | 11 (45)
Diarrhea (Gastrointestinal disorders) | 11 (46)
Dyspepsia (Gastrointestinal disorders) | 1 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 19 (71)
Vomiting (Gastrointestinal disorders) | 14 (45)
Edema limbs (General disorders) | 7 (11)
Fatigue (General disorders) | 24 (134)
Fever (General disorders) | 8 (14)
Malaise (General disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 14 (70)
Lymphocyte count increased (Investigations) | 3 (3)
Neutrophil count decreased (Investigations) | 17 (38)
Platelet count decreased (Investigations) | 18 (77)
White blood cell decreased (Investigations) | 12 (43)
Anorexia (Metabolism and nutrition disorders) | 10 (18)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 4 (37)
Peripheral sensory neuropathy (Nervous system disorders) | 17 (106)
Presyncope (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Personality change (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (33)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (26)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (22)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes